CLINICAL TRIAL: NCT04603898
Title: Oxalate Formation From Ascorbic Acid
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, John Knight, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-300005614; R01DK126774 (NIH)
Record Dates: First submitted 2020-10-21; First posted 2020-10-27 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Kidney Stone
Keywords: Oxalate; Calcium oxalate stones; Ascorbic Acid
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Controlled Dietary Study (Experimental): Subjects will consume a controlled diet (low in oxalate and ascorbic acid) for six days. After two days of equilibration, subjects will provide a blood sample and ingest an oral load of ascorbic acid (1 mg/kg) with breakfast on Day 3. The following day (Day 4), serial blood and urine collections will occur. On Days 5 through 7, subjects will complete a 24-hr urine collection and blood draw.
  Interventions: Dietary Supplement: Low Oxalate Diet; Dietary Supplement: Carbon-13 Ascorbic Acid Oral Load

INTERVENTIONS:
Dietary Supplement: Low Oxalate Diet — Subjects will be instructed to ingest a controlled diet low in oxalate for a total of 4 days
Dietary Supplement: Carbon-13 Ascorbic Acid Oral Load — Subjects will be instructed to ingest 1mg/kg of carbon-13 ascorbic acid at breakfast, 2 days after initiating the low oxalate controlled diet.

SUMMARY:
The purpose of this basic research study is to determine the contribution of endogenous ascorbic acid (AA) turnover to urinary oxalate excretion in both normal BMI and obese adult non-stone formers and calcium oxalate stone formers. The studies proposed will use diets of known nutrient composition, a stable isotope of ascorbic acid (13C6-AA) and mass spectrometric techniques to quantify ascorbic acid turnover to oxalate.

DETAILED DESCRIPTION:
The purpose of this basic research study is to determine the contribution of endogenous ascorbic acid (AA)turnover to urinary oxalate excretion in both normal BMI and obese adult non-stone formers and calcium oxalate stone formers. The studies proposed will use diets of known nutrient composition, a stable isotope of AA, 13C6-AA, and mass spectrometric techniques to quantify AA turnover to oxalate.

Adults (≥19 years) with and without a history of calcium oxalate kidney stone disease will be recruited from within the greater Birmingham area, and divided into normal BMI (BMI<25 kg/m2) and obese (BMI≥30 kg/m2) groups. Following consent, subjects will meet with a dietitian to ensure willingness to consume controlled diets, and provide fasted blood and 2 x 24 hour urine specimens to determine general health status and adequacy of 24-hour urine collections, respectively.

Eligible subjects will consume a low oxalate controlled diet for 6 days, which will involve 2 days of dietary equilibration followed by oral ingestion of 1 mg/kg carbon-13 AA with breakfast on day 3 and subsequent collection of 4 consecutive 24-hour urine specimens. After the carbon-13 AA load, subjects will return each morning to the Clinical Research Unit for a fasted blood draw, to drop off their 24-hour urine collection, and receive their prepared food. In addition, on day 4, 24 hours after ingesting carbon-13 AA, subjects will collect hourly urine and 1/2 hourly blood samples for 5 hours in the Clinical Research Unit.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* For stone formers: composition of most recent stone > 50% calcium oxalate, no uric acid component
* For stone formers: first time or recurrent calcium oxalate stone former with stone event within the prior 3 years
* Two 24-hour urine collections with urinary 24-hour creatinine excretion within 20% of appropriate ratio of creatinine (mg) / body weigh (kg) for gender
* Willingness to stop supplements (vitamins, Calcium (citrate or carbonate) and other minerals, herbal supplements, nutritional aids, probiotics) for 2 weeks before start and during study
* Willingness to not undertake vigorous exercise during the study
* Normal fasting blood Comprehensive Metabolic Panel (CMP)
* Willingness to ingest menus prepared in Clinical Research Unit at University of Alabama at Birmingham
* No food allergies or intolerance to any of the foods in study menus
* If on medications for stone prevention (e.g. thiazides, citrate supplementation excluding calcium citrate), they should have been on a stable dose regimen for at least 8 weeks prior to and during screening, with no changes in dosing anticipated during study protocol. If on allopurinol for stone prevention, stop it for 2 weeks prior to screening and this will not be administered during the study as it has anti-oxidant properties.

Exclusion Criteria:

* Diabetes
* Gout
* Hypertension
* Estimated Glomerular Filtration Rate (eGFR) less than 60ml/min/1.73m2
* Primary hyperoxaluria
* Nephrotic syndrome
* Enteric hyperoxaluria
* Renal tubular acidosis
* Primary hyperparathyroidism
* Liver disease
* Auto-immune disorder
* Neurogenic bladder
* Urinary diversion
* Bariatric surgery
* Active malignancy or treatment for malignancy within 12 months prior to screening
* Pregnancy
* Breastfeeding/nursing individuals
* Females of child bearing age who are not able to use an effective method of birth control during the study
* Mental/medical condition that is likely to impede successful study completion
* Illness including flu/common cold/fever 14 days before study and during study
* Diarrhea or other abnormal gastrointestinal event (e.g. abnormal bowel movements) 14 days before study or during study
* Abnormal fasting CMP

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Percent contribution of ascorbic acid (AA) to urinary oxalate excretion | Day 4
  On the last day (Day 4) of controlled diet and 24 hours following ingestion of an oral load of carbon-13 AA (1mg/kg), urine and blood will be collected and the levels of carbon 12 and carbon 13 AA and oxalate measured to determine the percent contribution of AA metabolism to urinary oxalate excretion for each subject.

CONTACTS AND LOCATIONS:
Overall Officials: John Knight, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No